CLINICAL TRIAL: NCT02132741
Title: Assessment of Retinal Vasculature Using Optical Coherence Tomography in Health, Hypertension & Chronic Kidney Disease.
Brief Title: Optical Coherence Tomography And NEphropathy: The OCTANE Study
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 14/SS/0069
Record Dates: First submitted 2014-04-29; First posted 2014-05-07 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2024-06

CONDITIONS: Health; Hypertension; Chronic Kidney Disease
Keywords: OCT; hypertension; CKD
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Treated hypertension: Patients on treatment for hypertension
- CKD-ESRD: Pre- & post haemodialysis
- Healthy individuals: Healthy volunteers
- Chronic kidney disease: Pre-dialysis CKD & those with a functional renal transplant
- Hypertension: Untreated

SUMMARY:
Patients with high blood pressure (hypertension) and chronic kidney disease are at an increased risk of developing heart disease and strokes. Part of this risk is due to changes in the structure and function of the blood vessels throughout the body. It is thought that reducing high blood pressure and treating chronic kidney disease improves the structure and function of blood vessels but information on this is limited. Optical coherence tomography (OCT) is a method of looking at the blood vessels at the back of the eye. It is a simple, quick and non-invasive test that you may have previously had during a visit to the optician. The purpose of the study is to ascertain whether OCT is able to detect changes in the eye's blood vessels in patients with hypertension and chronic kidney disease compared to healthy individuals and also to see if any differences seen improve with treatment.

DETAILED DESCRIPTION:
This project is an exploratory study, using enhanced depth imaging with the new SPECTRALIS OCT, designed to examine choroidal and microvascular retinal structure in patients with hypertension, chronic kidney disease (CKD), and in age and sex matched healthy controls. The study is non-invasive and takes only a few seconds to acquire these complex images. The Centre, where the images will be captured and where image analysis systems are located, is on the Royal Infirmary of Edinburgh (RIE) site close to the RIE outpatient clinics, making recruitment easy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-80
* Body mass index ≤35
* For those with hypertension: BP ≥140/90 or on treatment for hypertension
* For those with CKD: CKD as defined by the Kidney Diseases Quality Initiative guidelines

Exclusion Criteria:

* Subject is below the age of legal consent, or is mentally or legally incapacitated
* The subject has donated blood (450 ml) within the last 4 weeks
* Past or present drug or alcohol abuse including intravenous drug abuse at any time
* Participation in another clinical trial within 1 month
* Considered to be at high risk of HIV or hepatitis B
* Patients with known eye disease, or previous eye surgery, or refractive error greater than +/- 6 dioptres.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be recruited from a research database. CKD and patients with hypertension will be recruited from these respective clinics in secondary care.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-05-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Choroidal & retinal morphology | 2 weeks
  A composite measures outcome including:
  1. Sub-foveal choroidal thickness
  2. Choroidal volume
  3. Retinal vasculature morphology and optimality measurements (arteriolar thickness, branching coefficient and branching angle; fractal dimension, and venular tortuosity.)

SECONDARY OUTCOMES:
Neuro-retinal metrics | 2 weeks
  A composite measures outcome of neuro-retinal metrics (retinal thickness, retinal nerve fibre layer thickness)

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Dhaun, MD PhD, Principal Investigator — University of Edinburgh
Locations (1):
- University of Edinburgh, Edinburgh, Midlothian, United Kingdom

REFERENCES:
- [Derived] Balmforth C, van Bragt JJ, Ruijs T, Cameron JR, Kimmitt R, Moorhouse R, Czopek A, Hu MK, Gallacher PJ, Dear JW, Borooah S, MacIntyre IM, Pearson TM, Willox L, Talwar D, Tafflet M, Roubeix C, Sennlaub F, Chandran S, Dhillon B, Webb DJ, Dhaun N. Chorioretinal thinning in chronic kidney disease links to inflammation and endothelial dysfunction. JCI Insight. 2016 Dec 8;1(20):e89173. doi: 10.1172/jci.insight.89173. PMID 27942587